CLINICAL TRIAL: NCT02201901
Title: A Phase 3, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/GS-5816 Fixed-Dose Combination in Subjects With Chronic HCV Infection and Child-Pugh Class B Cirrhosis
Brief Title: Sofosbuvir/Velpatasvir Fixed-Dose Combination in Adults With Chronic HCV Infection and Child-Pugh Class B Cirrhosis
Acronym: ASTRAL-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-1137
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2016-10

CONDITIONS: Hepatitis C Virus Infection
Keywords: Sofosbuvir; Velpatasvir; SOF/VEL; GS-5816; Hepatitis C; HCV; Cirrhosis; CPT-B
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SOF/VEL 12 weeks (Experimental): Participants will receive SOF/VEL FDC for 12 weeks.
  Interventions: Drug: SOF/VEL
- SOF/VEL+RBV 12 weeks (Experimental): Participants will receive SOF/VEL FDC plus RBV for 12 weeks.
  Interventions: Drug: SOF/VEL; Drug: RBV
- SOF/VEL 24 weeks (Experimental): Participants will receive SOF/VEL FDC for 24 weeks.
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg tablets administered orally once daily
  Other Names: GS-7977/GS-5816; Epclusa®
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: SOF/VEL+RBV 12 weeks

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of sofosbuvir (SOF)/velpatasvir (VEL) fixed dose combination (FDC) with and without ribavirin (RBV) for 12 weeks and SOF/VEL FDC for 24 weeks in adults with chronic hepatitis C virus (HCV) infection and Child-Pugh-Turcotte (CPT) class B cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA > 10^4 IU/mL at screening
* Chronic HCV infection (≥ 6 months)
* Confirmed CPT class B (7-9) at screening

Exclusion Criteria:

* Current or prior history of solid organ transplantation, significant pulmonary disease, significant cardiac disease, or porphyria
* Inability to exclude hepatocellular carcinoma (HCC) by imaging within 6 months of baseline/Day 1
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Screening ECG with clinically significant abnormalities
* Prior exposure to SOF or any other nucleotide analogue HCV nonstructural protein 5B (NS5B) inhibitor or any HCV NS5A inhibitor
* Laboratory results outside of acceptable ranges at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anu M Osinusi, MD, MPH, Study Director — Gilead Sciences
Locations (44):
- United States (43):
  - Phoenix, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Pasadena, California
  - San Francisco, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Tampa, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Monroe, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Rochester, Minnesota
  - Jackson, Mississippi
  - St Louis, Missouri
  - Santa Fe, New Mexico
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Murray, Utah
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Background] Charlton MR, O'Leary JG, Bzowej NH, Muir AJ, Korenblat KM, Fenkel JM, et al. Sofosbuvir/Velapatasvir Fixed Dose Combination for the Treatment of HCV in Patients with Decompensated Liver Disease: The Phase 3 ASTRAL-4 Study. Hepatology 2015; 62 (6): 1387A-1388A.
- [Result] Curry MP, O'Leary JG, Bzowej N, Muir AJ, Korenblat KM, Fenkel JM, Reddy KR, Lawitz E, Flamm SL, Schiano T, Teperman L, Fontana R, Schiff E, Fried M, Doehle B, An D, McNally J, Osinusi A, Brainard DM, McHutchison JG, Brown RS Jr, Charlton M; ASTRAL-4 Investigators. Sofosbuvir and Velpatasvir for HCV in Patients with Decompensated Cirrhosis. N Engl J Med. 2015 Dec 31;373(27):2618-28. doi: 10.1056/NEJMoa1512614. Epub 2015 Nov 16. PMID 26569658
- [Result] Asselah T, Charlton M, Feld J, Foster GR, McNally J, Brainard DM, et al. The ASTRAL Studies: Evaluation of SOF/GS-5816 Single-Tablet Regimen for the Treatment of Genotype 1-6 HCV Infection [Poster P1332]. J Hepatol 2015; 62:S855-S6.
- [Derived] Younossi ZM, Stepanova M, Charlton M, Curry MP, O'Leary JG, Brown RS, Hunt S. Patient-reported outcomes with sofosbuvir and velpatasvir with or without ribavirin for hepatitis C virus-related decompensated cirrhosis: an exploratory analysis from the randomised, open-label ASTRAL-4 phase 3 trial. Lancet Gastroenterol Hepatol. 2016 Oct;1(2):122-132. doi: 10.1016/S2468-1253(16)30009-7. Epub 2016 Aug 3. PMID 28404069
- [Derived] Younossi ZM, Stepanova M, Feld J, Zeuzem S, Sulkowski M, Foster GR, Mangia A, Charlton M, O'Leary JG, Curry MP, Nader F, Henry L, Hunt S. Sofosbuvir and Velpatasvir Combination Improves Patient-reported Outcomes for Patients With HCV Infection, Without or With Compensated or Decompensated Cirrhosis. Clin Gastroenterol Hepatol. 2017 Mar;15(3):421-430.e6. doi: 10.1016/j.cgh.2016.10.037. Epub 2016 Nov 12. PMID 27847279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 47 study sites in the United States. The first participant was screened on 31 July 2014. The last study visit occurred on 25 November 2015.
Pre-assignment Details: 438 participants were screened.
Groups:
- SOF/VEL 12 Weeks (Group 1): SOF/VEL (Sofosbuvir/velpatasvir) (400/100 mg) fixed dose combination (FDC) tablet once daily for 12 weeks
- SOF/VEL+RBV 12 Weeks (Group 2): SOF/VEL (400/100 mg) FDC tablet + Ribavirin (RBV) tablets (1000 or 1200 mg/day divided twice daily) administered orally once daily for 12 weeks
- SOF/VEL 24 Weeks (Group 3): SOF/VEL (400/100 mg) FDC tablet once daily for 24 weeks
Period: Overall Study
Arm/Group | SOF/VEL 12 Weeks (Group 1) | SOF/VEL+RBV 12 Weeks (Group 2) | SOF/VEL 24 Weeks (Group 3)
Started | 90 | 88 | 90
Completed | 75 | 79 | 77
Not Completed | 15 | 9 | 13
Not completed — Randomized but never treated | 0 | 1 | 0
Not completed — Lack of Efficacy | 7 | 1 | 6
Not completed — Death | 3 | 3 | 3
Not completed — Lost to Follow-up | 2 | 3 | 2
Not completed — Withdrew Consent | 2 | 0 | 2
Not completed — Adverse Event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug.
Groups:
- SOF/VEL 24 Weeks ((Group 3): SOF/VEL (400/100 mg) FDC tablet once daily for 24 weeks
- Total: Total of all reporting groups
Arm/Group | SOF/VEL 12 Weeks (Group 1) | SOF/VEL+RBV 12 Weeks (Group 2) | SOF/VEL 24 Weeks ((Group 3) | Total
Number analyzed (Participants) | 90 | 87 | 90 | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (6.3) | 58 (6.9) | 58 (5.8) | 58 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 21 | 27 | 81
  Male | 57 | 66 | 63 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 13 | 13 | 39
  Not Hispanic or Latino | 77 | 74 | 77 | 228
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 6 | 5 | 6 | 17
  White | 79 | 79 | 81 | 239
  Asian | 3 | 0 | 2 | 5
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Native Hawaiian or Pacific Islander | 0 | 1 | 0 | 1
  Other | 2 | 1 | 0 | 3
  Not Disclosed | 0 | 0 | 1 | 1
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 31 | 42 | 45 | 118
  ≥ 800,000 IU/mL | 59 | 45 | 45 | 149
HCV RNA [Mean (Standard Deviation); unit: log 10 IU/mL] | 6.0 (0.54) | 5.8 (0.61) | 5.9 (0.63) | 5.9 (0.60)
HCV Genotype [Number; unit: participants]
  Genotype 1 | 68 | 68 | 71 | 207
  Genotype 2 | 4 | 4 | 4 | 12
  Genotype 3 | 14 | 13 | 12 | 39
  Genotype 4 | 4 | 2 | 2 | 8
  Genotype 6 | 0 | 0 | 1 | 1
IL28B [Number; unit: participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 20 | 22 | 20 | 62
    CT | 51 | 46 | 49 | 146
    TT | 19 | 19 | 19 | 57
    Missing | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: The Full Analysis Set (FAS): participants who were randomized into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL 12 Weeks (Group 1): SOF/VEL (400/100 mg) FDC tablet once daily for 12 weeks
- SOF/VEL+RBV 12 Weeks (Group 2): SOF/VEL (400/100 mg) FDC tablet + RBV tablets (1000 or 1200 mg/day divided twice daily) administered orally once daily for 12 weeks
Arm/Group | SOF/VEL 12 Weeks (Group 1) | SOF/VEL+RBV 12 Weeks (Group 2) | SOF/VEL 24 Weeks (Group 3)
Number analyzed (Participants) | 90 | 87 | 90
percentage of participants | 83.3 [74.0 to 90.4] | 94.3 [87.1 to 98.1] | 87.8 [79.2 to 93.7]
Statistical Analysis 1: Comparison: SOF/VEL 12 Weeks (Group 1); A sample size of 75 participants per treatment group would provide over 99% power to detect 40% improvement in SVR12 rate from the assumed spontaneous rate of 1% or less using a 2-sided exact 1-sample binomial test at significance level of 0.0167; Test type: Superiority or Other; p < 0.001, Binomial test; P-value is from the 2-sided exact 1-sample binomial test for the superiority of SOF/VEL 12 weeks (Group 1) over prespecified rate of 1%
Statistical Analysis 2: Comparison: SOF/VEL+RBV 12 Weeks (Group 2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Binomial test; P-value is from the 2-sided exact 1-sample binomial test for the superiority of SOF/VEL+RBV 12 weeks (Group 2) over prespecified rate of 1%
Statistical Analysis 3: Comparison: SOF/VEL 24 Weeks (Group 3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Binomial test; P-value is from the 2-sided exact 1-sample binomial test for the superiority of SOF/VEL 24 weeks (Group 3) over prespecified rate of 1%

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks (Group 1) | SOF/VEL+RBV 12 Weeks (Group 2) | SOF/VEL 24 Weeks (Group 3)
Number analyzed (Participants) | 90 | 87 | 90
percentage of participants | 1.1 | 16.1 | 4.4

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL+RBV 12 Weeks (Group 2): SOF/VEL (400/100mg) FDC tablet + RBV tablets (1000 or 1200 mg/day divided twice daily) administered orally once daily for 12 weeks
Arm/Group | SOF/VEL 12 Weeks (Group 1) | SOF/VEL+RBV 12 Weeks (Group 2) | SOF/VEL 24 Weeks (Group 3)
Number analyzed (Participants) | 90 | 87 | 90
percentage of participants
  SVR4 | 92.2 [84.6 to 96.8] | 95.4 [88.6 to 98.7] | 90.0 [81.9 to 95.3]
  SVR24 | 83.3 [74.0 to 90.4] | 94.3 [87.1 to 98.1] | 87.8 [79.2 to 93.7]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Weeks 1, 2, 4, 6, 8, 10, 12, 16, 20, and 24
Time Frame: Weeks 1, 2, 4, 6, 8, 10, 12, 16, 20, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks (Group 1) | SOF/VEL+RBV 12 Weeks (Group 2) | SOF/VEL 24 Weeks (Group 3)
Number analyzed (Participants) | 90 | 87 | 90
percentage of participants
  Wk 1(Group 1: N=90; Group 2: N=87; Group 3: N=90) | 2.2 | 14.9 | 11.1
  Wk 2 (Group 1: N=90; Group 2: N=87;Group 3: N=89) | 34.4 | 49.4 | 39.3
  Wk 4 (Group 1: N=90; Group 2: N=87; Group 3: N=89) | 81.1 | 80.5 | 91.0
  Wk 6(Group 1: N=89; Group 2: N=85; Group 3: N=88) | 98.9 | 97.6 | 98.9
  Wk 8(Group 1: N=89; Group 2: N=84; Group 3: N=87) | 98.9 | 98.8 | 100.0
  Wk 10(Group 1: N=89; Group 2: N=84; Group 3: N=87) | 100.0 | 98.8 | 100.0
  Wk 12(Group 1: N=89; Group 2: N=83; Group 3: N=87) | 100.0 | 98.8 | 97.7
  Wk 16(Group 1: N=0; Group 2: N=0; Group 3: N=86) | NA — Treatment for this group was only 12 weeks. | NA — Treatment for this group was only 12 weeks. | 97.7
  Wk 20(Group 1: N=0; Group 2: N=0;Group 3: N=84) | NA — Treatment for this group was only 12 weeks. | NA — Treatment for this group was only 12 weeks. | 100.0
  Wk 24(Group 1: N=0; Group 2: N=0; Group 3: N=84) | NA — Treatment for this group was only 12 weeks. | NA — Treatment for this group was only 12 weeks. | 100.0

5. Secondary Outcome: Change From Baseline in HCV RNA at Weeks 1, 2, 4, 6, 8, 10, 12, 16, 20, and 24
Time Frame: Baseline; Weeks 1, 2, 4, 6, 8, 10, 12, 16, 20, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL 12 Weeks (Group 1) | SOF/VEL+RBV 12 Weeks (Group 2) | SOF/VEL 24 Weeks (Group 3)
Number analyzed (Participants) | 90 | 87 | 90
log10 IU/mL
  Wk 1(Group 1: N=89; Group 2: N=83; Group 3: N=88) | -3.51 (0.652) | -3.63 (0.691) | -3.72 (0.680)
  Wk 2(Group 1: N=89; Group 2: N=87; Group 3: N=88) | -4.24 (0.677) | -4.17 (0.647) | -4.38 (0.669)
  Wk 4(Group 1: N=88; Group 2: N=86; Group 3: N=88) | -4.78 (0.549) | -4.58 (0.568) | -4.70 (0.613)
  Wk 6(Group 1: N=89; Group 2: N=85; Group 3: N=88) | -4.87 (0.536) | -4.68 (0.607) | -4.74 (0.630)
  Wk 8(Group 1: N=89; Group 2: N=83; Group 3: N=87) | -4.87 (0.536) | -4.68 (0.622) | -4.76 (0.613)
  Wk 10(Group 1: N=89; Group 2: N=84; Group 3, N=87) | -4.87 (0.536) | -4.67 (0.634) | -4.76 (0.613)
  Wk 12(Group 1: N=89; Group 2: N=82; Group 3: N=86) | -4.87 (0.536) | -4.68 (0.624) | -4.75 (0.618)
  Wk 16 (Group 1: N=0; Group 2: N=0; Group 3: N=85) | NA (NA) — Treatment for this group was 12 weeks only. | NA (NA) — Treatment for this group was 12 weeks only. | -4.76 (0.617)
  Wk 20 (Group 1: N=0; Group 2: N=0; Group 3: N =84) | NA (NA) — Treatment for this group was 12 weeks only. | NA (NA) — Treatment for this group was 12 weeks only. | -4.77 (0.613)
  Wk 24 (Group 1: N=0; Group 2: N=0; Group 3: N =84) | NA (NA) — Treatment for this group was 12 weeks only. | NA (NA) — Treatment for this group was 12 weeks only. | -4.77 (0.613)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as
  * On-treatment virologic failure
    * HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ, while on treatment,
    * > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment,
    * HCV RNA persistently ≥ LLOQ through 8 weeks of treatment (ie nonresponse)
  * Relapse
    * HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks (Group 1) | SOF/VEL+RBV 12 Weeks (Group 2) | SOF/VEL 24 Weeks (Group 3)
Number analyzed (Participants) | 90 | 87 | 90
percentage of participants | 12.2 [6.3 to 20.8] | 3.4 [0.7 to 9.7] | 8.9 [3.9 to 16.8]

7. Secondary Outcome: Percentage of Participants With a Decrease, No Change, or Increase Between Baseline and Posttreatment Week 24 in MELD Score
Description: Model for End-Stage Liver Disease (MELD) scores are used to assess prognosis and suitability for liver transplantation. Scores can range from 6 to 40; higher scores/increased scores indicate greater severity of disease.
Time Frame: Baseline to Posttreatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks (Group 1) | SOF/VEL+RBV 12 Weeks (Group 2) | SOF/VEL 24 Weeks (Group 3)
Number analyzed (Participants) | 69 | 75 | 69
percentage of participants
  Decrease (Improvement) | 55.1 | 49.3 | 50.7
  No Change | 20.3 | 25.3 | 21.7
  Increase (Worsening) | 24.6 | 25.3 | 27.5

8. Secondary Outcome: Percentage of Participants With a Decrease, No Change, or Increase Between Baseline and Posttreatment Week 24 in Child-Pugh-Turcotte (CPT) Score
Description: CPT scores grade the severity of cirrhosis and are used to determine the need for liver transplantation. Scores can range from 5 to 15; higher scores/increased scores indicate greater severity of disease.
Time Frame: Baseline to Posttreatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks (Group 1) | SOF/VEL+RBV 12 Weeks (Group 2) | SOF/VEL 24 Weeks (Group 3)
Number analyzed (Participants) | 69 | 75 | 69
percentage of participants
  Decrease (Improvement) | 44.9 | 53.3 | 63.8
  No Change | 43.5 | 37.3 | 27.5
  Increase (Worsening) | 11.6 | 9.3 | 8.7

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF/VEL 12 Weeks (Group 1) | SOF/VEL+RBV 12 Weeks (Group 2) | SOF/VEL 24 Weeks (Group 3)
Serious Adverse Events (participants affected / at risk) | 17/90 | 14/87 | 16/90
Other Adverse Events (participants affected / at risk) | 65/90 | 74/87 | 61/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL 12 Weeks (Group 1) (N=90) | SOF/VEL+RBV 12 Weeks (Group 2) (N=87) | SOF/VEL 24 Weeks (Group 3) (N=90)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bone abscess (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1 | 1
Infectious colitis (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 3 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 2 | 2 | 1
Seizure (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL 12 Weeks (Group 1) (N=90) | SOF/VEL+RBV 12 Weeks (Group 2) (N=87) | SOF/VEL 24 Weeks (Group 3) (N=90)
Anaemia (Blood and lymphatic system disorders) | 4 | 26 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 7 | 6 | 4
Ascites (Gastrointestinal disorders) | 5 | 4 | 0
Constipation (Gastrointestinal disorders) | 6 | 3 | 6
Diarrhoea (Gastrointestinal disorders) | 6 | 18 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 8
Nausea (Gastrointestinal disorders) | 20 | 22 | 18
Vomiting (Gastrointestinal disorders) | 7 | 5 | 6
Fatigue (General disorders) | 23 | 34 | 21
Oedema peripheral (General disorders) | 7 | 6 | 7
Pyrexia (General disorders) | 6 | 4 | 3
Nasopharyngitis (Infections and infestations) | 2 | 3 | 8
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 8
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 10 | 4
Headache (Nervous system disorders) | 23 | 18 | 17
Insomnia (Psychiatric disorders) | 9 | 12 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 5 | 7
Hypertension (Vascular disorders) | 3 | 5 | 0

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years